CLINICAL TRIAL: NCT06898073
Title: Effects of Dual-task Training During Curved Walking for Cognitive Function in Stroke Patients
Brief Title: Dual-task Training During Curved Walking in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH24-CT8-05
Record Dates: First submitted 2025-03-09; First posted 2025-03-27 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Stroke Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive tasks as the second task in addition to walking (Experimental)
  Interventions: Behavioral: cognitive dual-task group
- walking without performing a second task during the walking training (Other)
  Interventions: Behavioral: Single-task group

INTERVENTIONS:
Behavioral: cognitive dual-task group — Cognitive tasks as the second task in addition to walking
  Arms: Cognitive tasks as the second task in addition to walking
Behavioral: Single-task group — walking without performing a second task during the walking training
  Arms: walking without performing a second task during the walking training

SUMMARY:
The purpose of this study is to explore the effects of curved walking training under dual-task conditions on the cognitive function and walking ability of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. First-time unilateral stroke
2. Age between 40 and 80 years
3. Able to walk 10 meters continuously with or without the use of assistive devices
4. Capable of following instructions and performing simple arithmetic
5. Brunnstrom stage 3 or higher

Exclusion Criteria:

1. Other neurological disease or unstable medical conditions
2. Visual field defect
3. Mini-Mental State Examination (MMSE) <24 points
4. Pusher syndrome
5. Half-sided neglect
6. Expressive aphasia
7. Poorly controlled hypertension or cardiovascular disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | From baseline to the end of treatment at 3 weeks
  Mini-Mental State Examination (MMSE) includes items such as orientation, attention, memory, language, verbal comprehension, executive function, and construction ability. The maximum score is 30 points. A higher score indicates better cognitive function. One point is given for each correct answer. A total score below 24 suggests mild cognitive impairment, while a score below 16 indicates severe cognitive impairment.
Trail Making Test | From baseline to the end of treatment at 3 weeks
  The test consists of two parts, A and B. In part A, the participant is asked to connect a series of numbers in sequential order as quickly as possible. Part B includes both numbers and colors, where the participant must alternate between connecting the numbers and colors in order. The test records the time taken to complete the sequence and the number of errors made for scoring. If part B is not completed within 5 minutes, the test is stopped, and the highest score of 300 seconds is recorded. A lower score indicates faster completion time, suggesting better function.
Walking ability with different attention loads while turning - time | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a continuous curved path, without or with dual tasks. The time (seconds) taken to turn will be recorded using a stopwatch.
Walking ability with different attention loads while turning - numbers of steps | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a continuous curved path, without or with dual tasks. The numbers of steps taken to turn will be recorded using a counter.
Walking ability with different attention loads while turning - gait speed | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a continuous curved path, without or with dual tasks. Gait speed (m/s) will be recorded using the commercially available portable gait analysis system (Gait Up).
Walking ability with different attention loads while turning - step length | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a continuous curved path, without or with dual tasks. Step length (cm) during gait will be recorded and analyzed using the commercially available portable gait analysis system (Gait Up).
Walking ability with different attention loads while turning - step time | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a continuous curved path, without or with dual tasks. Step time (seconds) will be recorded and analyzed using the commercially available portable gait analysis system (Gait Up).
Walking ability with different attention loads while straight-line walking - time | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a straight-line path, without or with dual tasks. The time taken to turn will be recorded using a stopwatch.
Walking ability with different attention loads while straight-line walking - numbers of steps | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a straight-line path, without or with dual tasks. The numbers of steps taken to turn will be recorded using a counter.
Walking ability with different attention loads while straight-line walking - gait speed | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a straight-line path, without or with dual tasks. Gait speed will be recorded using the commercially available portable gait analysis system (Gait Up).
Walking ability with different attention loads while straight-line walking - step length | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a straight-line path, without or with dual tasks. Step length (cm) will be recorded using the commercially available portable gait analysis system (Gait Up).
Walking ability with different attention loads while straight-line walking - step time | From baseline to the end of treatment at 3 weeks
  The participant will be asked to walk 10 meters in a straight-line path, without or with dual tasks. Step time (second) will be recorded using the commercially available portable gait analysis system (Gait Up).
Timed up and go test | From baseline to the end of treatment at 3 weeks
  This test requires a 3-meter distance to be marked on the floor, with a chair placed at one end. The time which the participant stands up, walks forward to the 3-meter mark, turns around, walks back to the chair, and sits down again will be calculated and recorded.
Time taken to complete the Figure-of-Eight Walk test | From baseline to the end of treatment at 3 weeks
  The figure-eight walking test path includes both straight and turning paths. The participant will first be asked to stand between two traffic cones, spaced 5 feet apart. They will then be instructed to walk forward, turn around the first cone in their preferred direction, return to the starting point, and then turn around the second cone in the opposite direction before returning to the center. The time taken to complete the figure-eight walking test will be recorded.
Numbers of steps to complete the Figure-of-Eight Walk test | From baseline to the end of treatment at 3 weeks
  The figure-eight walking test path includes both straight and turning paths. The participant will first be asked to stand between two traffic cones, spaced 5 feet apart. They will then be instructed to walk forward, turn around the first cone in their preferred direction, return to the starting point, and then turn around the second cone in the opposite direction before returning to the center. Numbers of steps to complete the Figure-of-Eight Walk test will be recorded.

SECONDARY OUTCOMES:
Berg Balance Scale | From baseline to the end of treatment at 3 weeks
  This scale includes 14 test items. The scoring for each item ranges from 0 to 4. Generally, a score of 0 means the participant is completely unable to perform the test, while a score of 4 means the participant can complete the action within the specified time or achieve the maximum required distance or range of motion for the task. Each test item has a clear description of the scoring criteria. The total score is 56, and a higher score indicates better balance ability.
Activities-Specific Balance Confidence scale | From baseline to the end of treatment at 3 weeks
  This is a questionnaire that assesses the participant's level of self-confidence in maintaining balance in 16 situations commonly encountered in the community. Each of the 16 items is scored starting from 0, where 0 indicates no confidence, and scores increase in intervals of 10, with a maximum score of 100. A score of 100 represents complete confidence in maintaining balance.
Number of falls | From baseline to the end of treatment at 3 weeks
  The number of falls experienced by the participant in the past year will first be recorded. The participant will then be provided with a fall diary to track the number of falls during the one-year follow-up period after the assessment. In this study, a fall is defined as when the individual unintentionally falls to the ground, floor, or another lower level position. Each month, a follow-up phone call will be made to ensure the participant is recording the fall count as required.

CONTACTS AND LOCATIONS:
Locations (1):
- Fooyin University, Kaohsiung City, Taiwan